CLINICAL TRIAL: NCT01290120
Title: Multicentre Study to Optimize Therapy of Burkitt's Leukemia (B-ALL) and Non-Hodgkin Lymphoma
Brief Title: Chemotherapy Plus Rituximab Combination for Adult Lymphoblastic Leukemia (B-ALL) and Burkitt's Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northern Italy Leukemia Group (Other)
Responsible Party: Principal Investigator, DR RENATO BASSAN, MD, Northern Italy Leukemia Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NILG 2009-012950-19
Record Dates: First submitted 2011-02-02; First posted 2011-02-04 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Burkitt Lymphoma; B-ALL
Keywords: Burkitt Lymphoma; B-ALL; Adult patients
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Rituximab; Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Chemotherapy-Rituximab combination — Short cycles of high-dose and conventional chemotherapy in combination with rituximab, followed by local radiotherapy in the case of initial mediastinal or central nervous system (CNS) involvement or a residual tumor after chemotherapy. Used drugs are rituximab,cyclophosphamide, prednisone, dexamethasone, vincristine, methotrexate, iphosphamide, teniposide, etoposide, dexamethasone, cytarabine,adriamycin, vincristine, vindesine.
  Other Names: Mabthera; Rituxan; Endoxan; Aracytin; Doxorubicin; Vepesid

SUMMARY:
The study was set up to assess the efficacy and tolerability of a chemotherapy-immunotherapy combination programme originally introduced by GMALL (the German cooperative group for adult acute lymphoblastic leukemia)in 2002, to improve remission rate, overall and disease-free survival rates of adult patients with Burkitt's leukemia and lymphoma.

The therapy includes a maximum of six chemotherapy courses (two with high doses of methotrexate and cytarabine) plus anti-CD20 antibody (Rituximab, up to 8 total doses), supplemented by local radiation therapy in the case of initial mediastinal or central nervous system (CNS) involvement or a residual tumor after chemotherapy.

DETAILED DESCRIPTION:
Cycle A1: prednisone-cyclophosphamide pre-phase (5 days), Rituximab on day 0, chemotherapy on days 1-5 (dexamethasone, iphosphamide, vincristine, high-dose methotrexate, triple intrathecal therapy).

Cycle B1: Rituximab on day 0, chemotherapy on days 1-5 (dexamethasone, vincristine, cyclophosphamide, high-dose methotrexate, adriamycin, triple intrathecal therapy) Cycle C1: Rituximab on day 0, chemotherapy on days 1-5 (dexamethasone, vindesine, high-dose methotrexate, etoposide, high-dose cytarabine).

Cycle A2: like cycle A1, without pre-phase. Cycle B2: like cycle B1. Cycle C2: like cycle C1. Cycle C2 is followed by two additional Rituximab injections.

Notes:

1. patients with stage I-II disease without mediastinal tumor or extranodal involvement receive only the first 4 cycles (A1 to A2).
2. patients aged >55 years do not receive cycles C (sequence: A1, B1, A2, B2, A3, B3 or A1, B1, A2, B2 if limited stage, with reduced-dose methotrexate).

ELIGIBILITY:
Inclusion Criteria:

* Burkitt's leukemia or lymphoma (new diagnosis)
* Written informed consent
* Age > 15 years

Exclusion Criteria:

* pre-treated Burkitt's leukemia or lymphoma
* psychiatric disorders
* active second malignancy
* pregnancy
* absence of patient's written informed consent
* participation in other studies that interfere with the study therapy

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2002-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Percentage of patients alive without disease at 5 years from date of diagnosis

SECONDARY OUTCOMES:
Disease free survival | 5 years
  Percentage of patients alive without disease at 5 years from date of remission
Cumulative incidence of relapse | 5 years
  Percentage of relapsed patients at 5 years from date of remission
Complete remission rate | Up to 24 weeks
  Percentage of patients achieving complete remission after the first two treatment cycles (defining the early response rate), and then confirmed to remain in complete remission at end of the six chemotherapy blocks. Re-staging procedures include physical examination, blood counts and biochemistry, bone marrow examination , and instrumental tests as appropriate (ultrasound scans, computed tomography, nuclear magnetic resonance, positron emission tomography)depending on clinical presentation of individual subjects.
Toxicity | 1 year
  Percentage of patients who develop early and late therapy-related toxic side effects (including death in complete remision). Toxicity is defined according to the Common Toxicity Criteria scale (NCI), graded I-IV and referring to both hematological and extrahematologic toxicity. Early toxicity is registered during the first two chemotherapy cycles, and late toxicity following completion of therapy and up to 1 year from diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Renato Bassan, MD, Principal Investigator — USC Ematologia Ospedali Riuniti di Bergamo
Locations (12):
- Italy (12):
  - Divisione di Ematologia e TMO, Ospedale San Maurizio, Bolzano, (bz)
  - Ematologia e centro TMO - Ospedale Armando Businco, Cagliari, (ca)
  - S.C. Ematologia - Azienda Ospedaliera S. Croce e Carle, Cuneo, (cn)
  - Onco-Ematologia - Ospedale Civile, Noale, (ve)
  - Dipartimento di Ematologia e Medicina Trasfusionale - Azienda Osp. Nazionale Santi Antonio e Biagio e Cesare Arrigo, Alessandria, AL
  - USC Ematologia Ospedali Riuniti di Bergamo, Bergamo, BG
  - Divisione Ematologia Spedali Civili, Brescia, BS
  - Ematologia - AOU Careggi, Florence, FI
  - Ematologia e TMO - Ospedale San Raffaele, Milan, MI
  - Ematologia - TMO - Ospedale San Gerardo, Monza, MI
  - Ematologia Ospedale San Bortolo, Vicenza, VI
  - USC Ematologia Ospedali Riuniti di Bergamo, Bergamo

REFERENCES:
- [Derived] Intermesoli T, Rambaldi A, Rossi G, Delaini F, Romani C, Pogliani EM, Pagani C, Angelucci E, Terruzzi E, Levis A, Cassibba V, Mattei D, Gianfaldoni G, Scattolin AM, Di Bona E, Oldani E, Parolini M, Gokbuget N, Bassan R. High cure rates in Burkitt lymphoma and leukemia: a Northern Italy Leukemia Group study of the German short intensive rituximab-chemotherapy program. Haematologica. 2013 Nov;98(11):1718-25. doi: 10.3324/haematol.2013.086827. Epub 2013 Jun 10. PMID 23753030